CLINICAL TRIAL: NCT07361523
Title: Using Near-Infrared Spectroscopy Devices to Assess Myocardial and Visceral Perfusion During Complex Congenital Cardiac Surgery
Status: Not yet recruiting | Type: Observational
Sponsor: Boston Children's Hospital (Other)
Collaborators: ViOptix Canada (Industry)
Responsible Party: Principal Investigator, Sitaram Emani, Principal Investigator (PI), Boston Children's Hospital
Other Study IDs: IRB-P00052229
Record Dates: First submitted 2025-12-01; First posted 2026-01-23 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Congenital Heart Disease
MeSH Terms: conditions — Heart Defects, Congenital

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (1):
- IntraOx Device Patients: Pediatric patients undergoing congenital heart surgery with risk for myocardial or peripheral ischemia with use of IntraOx device intraoperatively to assess myocardial and visceral perfusion at 4 different time points
  Interventions: Device: Tissue oximeter (IntraOx)

INTERVENTIONS:
Device: Tissue oximeter (IntraOx) — The Intra.Ox device will be used to measure %StO2 readings taken at different time points during the surgery, including: (1) prior to bypass when the heart is being perfused by the coronary arteries, (2) after the patient is placed on cardiopulmonary bypass (CPB) but prior to placing a cross-clamp, (3) after placing a cross-clamp when the heart is not being perfused by CPB, and (4) after the patient is taken off CPB and the heart is re-perfusing. These readings will not impact the surgical management of the patient, and the congenital heart surgery will be carried out per standard of care according to the judgement of the surgeon.

SUMMARY:
The use of near infrared spectroscopy (NIRS) is a technique that has recently been incorporated by several other surgical specialties to measure tissue perfusion, such as in plastic surgery to allow for earlier detection of free flap vascular compromise in the postoperative monitoring protocol, with promising outcomes. IntraOx is a handheld oximeter that uses NIRS to measure tissue oxygen saturation and that has been used as an alternative to indocyanine green (ICG) to assess bowel perfusion in colorectal anastomotic cases. IntraOx is a promising technology that is also sterile and easy to use that can be incorporated into congenital heart surgery procedures to evaluate myocardial perfusion in a time sensitive manner. This technology could also be used on the liver to assess systemic perfusion as another indicator of cardiac function, in conjunction with the intraoperative transesophageal echocardiography (TEE). This could provide more concrete data about not only myocardial perfusion, but systemic perfusion as well. This data could be critical to help surgeons make surgical decisions and may help to improve patient outcomes.

This will be a prospective review of the use of the Intra.Ox device during cardiac surgery at different timepoints during the procedure to assess perfusion. This device is FDA-approved for use in adults but not approved for use in children and will be investigational in children.

The primary objective of this study is to test whether the Intra.Ox (Vioptix Inc.) using near-infrared spectroscopy to measure tissue oxygen saturation can be used to evaluate myocardial and visceral perfusion at different time points during complex congenital heart surgery, and particularly those involving coronary artery manipulation such as patients undergoing arterial switch operations or stage 1 palliation for hypoplastic left heart syndrome. The investigators would also use this device on the liver to assess systemic perfusion. The secondary objective is to evaluate whether the investigators would be able to use the information from the Intra.Ox device to make clinical decisions that can improve patient outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 1 year of age undergoing congenital heart surgery at Boston Children's Hospital are all eligible for participation in this study.
* All subjects undergoing congenital heart surgery at Boston Children's Hospital will be screened for inclusion in this study. Screening will prioritize identifying patients with concern for decreased myocardial and peripheral perfusion for any reason, as designated by Dr. Sitaram Emani's clinical judgement.
* Eligibility will be reviewed in advance by screening upcoming surgical procedures. All patients over 1 year of age will be eligible for participation in this study and screened for inclusion. Any patient at risk for malperfusion during bypass (e.g. Fontans, biventricular repair, long cross-clamp times, etc.) will be identified ahead of time and prioritized for inclusion in the study.

Exclusion Criteria:

* Any records flagged for "research opt out."
* Neonates and children undergoing surgery less than 1 year of age

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients over 1 year of age undergoing congenital heart surgery at Boston Children's Hospital identified by the PI and the study coordinator to have concern for decreased myocardial and peripheral perfusion for any reason. This may include, but will not be limited to, patients with history of myocardial ischemia, surgical procedures on the coronary arteries or operating near the coronary arteries that may impact myocardial perfusion, surgical procedures that may impact systemic perfusion, patients with history of coronary artery disease, patients with history of angina, patients with history of rheumatic disease that may impact perfusion, and patients with previous history of poor ventricular function, arrhythmia, or other complications following cardiopulmonary bypass.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Oxygen saturation | Day 0 ("baseline") up to 2 weeks post-operation
  Oxygen saturation levels measured from: pulse oximetry, tissue oximeter, arterial blood gases, and venous blood gases in units of %
Liver function test: ALP | Day 0 ("baseline") up to 2 weeks post-operation
  Post-operative liver function tests: Alkaline Phosphatase (ALP) in units of International Units per liter (U/L or IU/L) as a measure of the effects of systemic perfusion
Liver Function Test: AST | Day 0 ("baseline") up to 2 weeks post-operation
  Post-operative liver function test: AST (Aspartate Aminotransferase) in units of International Units per liter (U/L or IU/L) as a measure of the effects of systemic perfusion
Liver function Test: ALT | Day 0 ("baseline") up to 2 weeks post-operation
  Post-operative liver function test: ALT (Alanine Transaminase) in units of International Units per liter (U/L or IU/L) as a measure of the effects of systemic perfusion
Cardiac function | Day 0 ("baseline") up to 2 weeks post-operation
  Measuring cardiac function as measured by ejection fraction (in %) in post-operative echocardiogram results.
Kidney function | Day 0 ("baseline") up to 2 weeks post-operation
  Laboratory values of BUN and Creatinine (Cr) in units of mg/dL as a measurement of kidney function and perfusion
Mortality and major complications | Day 0 ("baseline") up to 2 weeks post-operation
  Major complications as defined by the STS and Congenital Heart Surgeons Society including renal failure requiring dialysis, permanent neurologic deficit, pacemaker, paralyzed diaphragm, mechanical circulatory support, and unplanned reintervention. This will be recorded as one outcome (whether or not a patient had mortality and major complications) and not measuring multiple multiple assessments; it is a quantitative assessment of whether or not a patient encountered one of the major complications or mortality as defined above. There are no units of measure.
Lactate | Day 0 ("baseline") up to 2 weeks post-operation
  Lactate levels in mmol/L as measurement for tissue perfusion.
pH | Day 0 ("baseline") up to 2 weeks post-operation
  pH from arterial blood gas and venous blood gas to measure blood acidity/alkalinity.
Blood gas: PaO2 | Day 0 ("baseline") up to 2 weeks post-operation
  PaO2 (partial pressures of oxygen) in mmHg from arterial and venous blood gas blood tests
Blood Gas: PaCO2 | Day 0 ("baseline") up to 2 weeks post-operation
  PaCO2 (partial pressures of carbon dioxide) in mmHg from arterial and venous blood gas blood tests
Bicarbonate | Day 0 ("baseline") up to 2 weeks post-operation
  Bicarbonate values from arterial and venous blood gas in units of mmol/L. This is one outcome measure that will be recorded, not multiple assessments with different units of measure. Bicarbonate values will be recorded from two different blood gas sources in mmol/L.
Echocardiography qualitative descriptions | Day 0 ("baseline") up to 2 weeks post-operation
  Measurement and recording of qualitative written report from cardiologist interpretation of echocardiography, specifically assessing for reports of 1) valvular dysfunction (regurgitation or stenosis), 2) myocardial dysfunction, hypokinesis, filling defects, etc. or 3) any other abnormalities written in qualitative report relating to cardiac function
Lactate | Day 0 ("baseline") up to 2 weeks post-operation
  Lactate levels in mmol/L as measurement for tissue perfusion

SECONDARY OUTCOMES:
Intensive care unit length of stay | Day 0 ("baseline") up to 2 weeks post-operation
  Intensive care unit length of stay in days
Hospital length of stay | Day 0 ("baseline") up to 2 weeks post-operation
  Hospital length of stay of stay in days
Liver function tests: bilirubin | Day 0 ("baseline") up to 2 weeks post-operation
  Measurements of bilirubin in units of mg/dL to assess liver function as indicator of tissue perfusion
Liver function test: protein | Day 0 ("baseline") up to 2 weeks post-operation
  Total protein in g/dL as measure of liver function
Liver function test: albumin | Day 0 ("baseline") up to 2 weeks post-operation
  Albumin in g/dL as measure of liver function
Electrolytes: sodium | Day 0 ("baseline") up to 2 weeks post-operation
  Basic metabolic panel laboratory value measuring sodium in units of mEq/L
Electrolytes: potassium | Day 0 ("baseline") up to 2 weeks post-operation
  Basic metabolic panel laboratory values measuring potassium in units of mEq/L
Electrolytes: chloride | Day 0 ("baseline") up to 2 weeks post-operation
  Basic metabolic panel laboratory values measuring chloride in units of mEq/L
Electrolytes: CO2 | Day 0 ("baseline") up to 2 weeks post-operation
  Basic metabolic panel laboratory values measuring CO2 in units of mEq/L
Basic metabolic panel: glucose | Day 0 ("baseline") up to 2 weeks post-operation
  Basic metabolic panel glucose levels in units of mg/dL
Basic metabolic panel: calcium | Day 0 ("baseline") up to 2 weeks post-operation
  Basic metabolic panel calcium levels in units of mg/dL
Aortic valve diameter | Day 0 ("baseline") up to 2 weeks post-operation
  Aortic heart valve annulus diameters measured in mm
Mitral valve diameter | Day 0 ("baseline") up to 2 weeks post-operation
  Mitral valve annulus diameters measured in mm
Pulmonary valve diameter | Day 0 ("baseline") up to 2 weeks post-operation
  Pulmonary valve annulus diameters measured in mm
Tricuspid valve diameter | Day 0 ("baseline") up to 2 weeks post-operation
  Tricuspid valve annulus diameters measured in mm
Heart valve pressure gradient: aortic valve | Day 0 ("baseline") up to 2 weeks post-operation
  Pressure gradients across aortic valve measured on echocardiography measured in mmHg
Heart valve pressure gradient: mitral valve | Day 0 ("baseline") up to 2 weeks post-operation
  Pressure gradients across mitral valve measured on echocardiography measured in mmHg
Heart valve pressure gradient: tricuspid valve | Day 0 ("baseline") up to 2 weeks post-operation
  Pressure gradients across tricuspid valve measured on echocardiography measured in mmHg
Heart valve pressure gradient: pulmonic valve | Day 0 ("baseline") up to 2 weeks post-operation
  Pressure gradients across pulmonic valve measured on echocardiography measured in mmHg

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pasquali SK, Shahian DM, O'Brien SM, Jacobs ML, Gaynor JW, Romano JC, Gaies MG, Hill KD, Mayer JE, Jacobs JP. Development of a Congenital Heart Surgery Composite Quality Metric: Part 1-Conceptual Framework. Ann Thorac Surg. 2019 Feb;107(2):583-589. doi: 10.1016/j.athoracsur.2018.07.037. Epub 2018 Sep 15. PMID 30227127
- [Background] Jacobs JP, Jacobs ML, Austin EH 3rd, Mavroudis C, Pasquali SK, Lacour-Gayet FG, Tchervenkov CI, Walters H 3rd, Bacha EA, Nido PJ, Fraser CD, Gaynor JW, Hirsch JC, Morales DL, Pourmoghadam KK, Tweddell JS, Prager RL, Mayer JE. Quality measures for congenital and pediatric cardiac surgery. World J Pediatr Congenit Heart Surg. 2012 Jan 1;3(1):32-47. doi: 10.1177/2150135111426732. PMID 23804682
- [Background] Koolen PGL, Vargas CR, Ho OA, Ibrahim AMS, Ricci JA, Tobias AM, Winters HAH, Lin SJ, Lee BT. Does Increased Experience with Tissue Oximetry Monitoring in Microsurgical Breast Reconstruction Lead to Decreased Flap Loss? The Learning Effect. Plast Reconstr Surg. 2016 Apr;137(4):1093-1101. doi: 10.1097/01.prs.0000481071.59025.82. PMID 27018663
- [Background] Oskarsson G, Pesonen E, Munkhammar P, Sandstrom S, Jogi P. Normal coronary flow reserve after arterial switch operation for transposition of the great arteries: an intracoronary Doppler guidewire study. Circulation. 2002 Sep 24;106(13):1696-702. doi: 10.1161/01.cir.0000030937.27602.bd. PMID 12270865
- [Background] Yates RW, Marsden PK, Badawi RD, Cronin BF, Anderson DR, Tynan MJ, Maisey MN, Baker EJ. Evaluation of myocardial perfusion using positron emission tomography in infants following a neonatal arterial switch operation. Pediatr Cardiol. 2000 Mar-Apr;21(2):111-8. doi: 10.1007/s002469910015. PMID 10754077
- [Background] Noel CV, Krishnamurthy R, Masand P, Moffett B, Schlingmann T, Cheong BY, Krishnamurthy R. Myocardial Stress Perfusion MRI: Experience in Pediatric and Young-Adult Patients Following Arterial Switch Operation Utilizing Regadenoson. Pediatr Cardiol. 2018 Aug;39(6):1249-1257. doi: 10.1007/s00246-018-1890-z. Epub 2018 May 10. PMID 29748700
- [Background] Sherwinter D, Chandler P, Martz J. The use of tissue oxygen measurements compared to indocyanine green imaging for the assessment of intraoperative tissue viability of human bowel. Surg Endosc. 2022 Mar;36(3):2192-2196. doi: 10.1007/s00464-021-08737-y. Epub 2021 Sep 22. PMID 34550436
- [Background] Khavanin N, Darrach H, Kraenzlin F, Yesantharao PS, Sacks JM. The Intra.Ox Near-Infrared Spectrometer Measures Variations in Flap Oxygenation That Correlate to Flap Necrosis in a Preclinical Rodent Model. Plast Reconstr Surg. 2021 May 1;147(5):1097-1104. doi: 10.1097/PRS.0000000000007894. PMID 33835088
- [Background] Gonzalez-Jacobo A, Chandler P, Martz J, Sherwinter D. Tissue Oximetry as a Potential Alternative to Indocyanine Green (ICG) Perfusion Assessment in Colorectal Anastomotic Cases. Surg Laparosc Endosc Percutan Tech. 2023 Apr 1;33(2):207-210. doi: 10.1097/SLE.0000000000001161. PMID 36971520
- [Background] Khavanin N, Almaazmi H, Darrach H, Kraenzlin F, Safar B, Sacks JM. Comparison of the ViOptix Intra.Ox Near Infrared Tissue Spectrometer and Indocyanine Green Angiography in a Porcine Bowel Model. J Reconstr Microsurg. 2020 Jul;36(6):426-431. doi: 10.1055/s-0040-1702163. Epub 2020 Feb 23. PMID 32088921
- [Background] Nguyen MB, Zhang N, Baranger J, Aguet J, Friedberg MK, Barron DJ, Honjo O, Mertens LL, Villemain O. Ultrafast Power Doppler for Detecting Intraoperative Myocardial Perfusion in Infants With Critical Congenital Heart Disease. JACC Adv. 2023 Apr 12;2(3):100290. doi: 10.1016/j.jacadv.2023.100290. eCollection 2023 May. No abstract available. PMID 38939593
- [Background] Said SM, Marey G, Hiremath G. Intraoperative fluorescence with indocyanine green in congenital cardiac surgery: Potential applications of a novel technology. JTCVS Tech. 2021 Feb 25;8:144-155. doi: 10.1016/j.xjtc.2021.02.026. eCollection 2021 Aug. PMID 34401838
- [Background] Goldman ME, Mindich BP. Intraoperative cardioplegic contrast echocardiography for assessing myocardial perfusion during open heart surgery. J Am Coll Cardiol. 1984 Nov;4(5):1029-34. doi: 10.1016/s0735-1097(84)80067-4. PMID 6333444
- [Background] Cyran SE, Kimball TR, Meyer RA, Bailey WW, Lowe E, Balisteri WF, Kaplan S. Efficacy of intraoperative transesophageal echocardiography in children with congenital heart disease. Am J Cardiol. 1989 Mar 1;63(9):594-8. doi: 10.1016/0002-9149(89)90905-3. PMID 2919563
- [Background] Nguyen MB, Zhang N, Mertens LL, Barron D, Honjo O, Venet M, Baranger J, Villemain O. Noninvasive assessment of myocardial perfusion using ultrafast ultrasound: clinical study for congenital heart disease. Eur Heart J Imaging Methods Pract. 2025 Jan 16;3(1):qyaf007. doi: 10.1093/ehjimp/qyaf007. eCollection 2025 Jan. PMID 39974276
- [Background] Congenital Heart Defects: What are Congenital Heart Defects? (2022). https://www.nhlbi.nih.gov/health/congenital-heart-defects.
- [Background] Singh Y, Lakshminrusimha S. Perinatal Cardiovascular Physiology and Recognition of Critical Congenital Heart Defects. Clin Perinatol. 2021 Aug;48(3):573-594. doi: 10.1016/j.clp.2021.05.008. PMID 34353581